CLINICAL TRIAL: NCT00746928
Title: Cardiovascular Consequences of Intermittent Hypoxia in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: TAMISIER Renaud, University Hospital, Grenoble
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 05-CHUG-23
Record Dates: First submitted 2008-09-01; First posted 2008-09-04 (Estimated); Last update posted 2008-09-04 (Estimated); Status verified 2008-09

CONDITIONS: Sleep Apnea Syndrome
Keywords: Blood pressure; Hypertension; sympathetic control; chemosensitivity; baroreflex
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Chronic Intermittent Hypoxia — Chronic Intermittent Hypoxia mimicking the CIH undergone by patients suffering from Sleep Apnea Syndrome, is applied to Healthy subject during 8 hours a day (nights) for a 14 days period. The cycle of intermittent Hypoxia is 30 drop in SaO2 per hours with a 10% decrease in SaO2.

SUMMARY:
The study is a prospective field evaluation to assess the effects of the chronic Intermittent Hypoxia exposure in 12 healthy humans.

Precisely, the study was designed to :

Set up a new model of Chronic Intermittent Hypoxia (CIH) applied to healthy human. This CIH is mimicking the CIH undergone by patients suffering from Sleep Apnea Syndrome.

Evaluate the cardiovascular effect of CIH. Neuronal and humoral sympathetic control, blood pressure control, vascular resistance.

Evaluate the Sleep quality, the ventilation under exposure and the long terms effect on ventilation control of CIH (central and peripheral chemoreflex).

Investigates the biological aspects of CIH exposure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Any history or significant medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-09; Primary Completion 2007-07 (Actual); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Two Weeks

SECONDARY OUTCOMES:
Neuronal and humoral sympathetic control and vascular resistance. | Two weeks
Sleep quality | Two Weeks
The ventilation under exposure and the long terms effect on ventilation control of CIH (central and peripheral chemoreflex) | two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Tamisier, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Pulmonary Function and sleep Lab, CHU Grenoble, Grenoble, France